CLINICAL TRIAL: NCT05420701
Title: A Study on Outcomes of Surgical and Percutaneous Left Atrial Appendage Closure
Brief Title: Surgical vs Percutaneous LAAO
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Chinese University of Hong Kong (Other)
Responsible Party: Principal Investigator, Professor Bryan Ping Yen YAN, Professor, Chinese University of Hong Kong
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2022.164
Record Dates: First submitted 2022-06-12; First posted 2022-06-15 (Actual); Last update posted 2022-09-21 (Actual); Status verified 2022-09

CONDITIONS: Atrial Fibrillation
Keywords: Left Atrial Appendage Closure; Left Atrial Appendage Occlusion
MeSH Terms: conditions — Atrial Fibrillation

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Left Atrial Appendage Occlusion (No Intervention)
- Left Atrial Appendage Closure, (Active Comparator)
  Interventions: Procedure: TEE

INTERVENTIONS:
Procedure: TEE — Patients in the surgical arm (LAAC) will be arranged to do TEE, which is not considered standard of care.
  Arms: Left Atrial Appendage Closure,

SUMMARY:
Atrial fibrillation is the most common cardiac arrythmia globally. Its prevalence ranges between 2-4% worldwide. It is associated with significant morbidity and mortality. One of the main concerns of AF is the risk of thromboembolism, which can result in debilitating or detrimental stroke. The gold standard for preventing AF stroke is long term oral anticoagulation in the form of warfarin or NOAC1,2.

Around 50% of patients who need anticoagulation are not on any form tablets and about 5% of patients who are not anticoagulated developed stroke. Some patients could not take anticoagulation because of high risk of bleeding, and this result in challenges within this cohort of patients. The left atrial appendage (LAA) is believed to be the main source of embolic in atrial fibrillation. The LAA is an anterolateral structure which is the smallest part of the left atrium. It originates anterior from the left pulmonary vein ostium. More than 90% of thromboembolic events happened in the LAA of non-rheumatic patients whereas only 57% of thrombi in rheumatic mitral valve disease3. This suggests that occluding the LAA is more beneficial in the non-valvular AF patients. Incomplete LAA closure is associated with a higher occurrence of thromboembolism. The growing evidence of LAA occlusion has been emerged. Percutaneous LAA Occlusion (LAAO) has been suggested that it may be considered for stroke prevention in patients with atrial fibrillation and contraindication for long term anticoagulation (class IIB, level B)1,2. This recommendation is based on the randomized controlled trials to show that percutaneous devices are non-inferior to oral anticoagulation in terms of preventing stroke in AF patients.

Surgical LAA clip occlusion (LAAC) has emerged as a potential method to isolate LAA to prevent thromboembolism. The recent LAAOS III trial shows that the risk of ischemic stroke or systemic embolism was lower with concomitant left atrial appendage occlusion performed during the surgery than without it, most of whom continued to receive ongoing anticoagulant therapy4. This reinforced the mechanistic value of occluding the LAA in prevention of stroke. However, the efficacy of isolated LAAC without anticoagulation is uncertain. Besides, as this surgical clip occlusion is frequently performed together with other concomitant cardiac surgery, post evaluation in the form of imaging is lacking. Our study aims to study the imaging follow-up result and clinical efficacy of surgical and percutaneous left atrial appendage closure.

ELIGIBILITY:
Inclusion Criteria:

* Atrial fibrillation diagnosis
* Underwent LAA clip (Atriclip) or left atrial appendage occlusion with CHADVASC >=2

Exclusion Criteria:

* Subject not required anticoagulation due to low CHADVASC
* Mechanical valve replacement
* Tissue mitral valve replacement or tissue aortic valve replacement with underlying chronic rheumatic heart disease

Min Age: 19 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 260 (Estimated)
Dates: Start 2022-10 (Estimated); Primary Completion 2026-12-31 (Estimated); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
occlusion result | around 1 year post procedure
  to compare the occlusion result of LAAC vs LAAO by transoesophageal echocardiogram.

IPD SHARING:
Plan to Share IPD: Undecided